CLINICAL TRIAL: NCT02012374
Title: Overcoming Learned Non-Use in Chronic Aphasia: Behavioral, fMRI and QoL Outcomes
Brief Title: Overcoming Learned Non-Use in Chronic Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-1065
Record Dates: First submitted 2013-02-12; First posted 2013-12-16 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Stroke-induced Aphasia
Keywords: aphasia; anomia; speech therapy; rehabilitation; neuroplasticity; fMRI; quality of life
MeSH Terms: conditions — Aphasia; Anomia; Communication Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Language Action Therapy ("constrained") (Experimental): Following a phase of baseline pre-treatment testing, speech therapy sessions take place 5 days/week for 3 hours per session during two consecutive weeks. Spoken responses are explicitly modeled and encouraged during therapy. Following the intensive 2-week treatment, participants are trained in using individualized home practice programs on iPads. They practice approximately daily for six months, checking in weekly with an SLP via videoconferencing software and return for probes monthly. Six months post-treatment testing will take place following completion of the home practice phase and again at 12 months post-treatment.
  Interventions: Behavioral: Intensive Language Action Therapy
- Unconstrained Intensive Language Action Therapy (Experimental): Following a phase of baseline pre-treatment testing, speech therapy sessions take place 5 days/week for 3 hours per session during two consecutive weeks. All communicative responses are encouraged during therapy. Following the intensive 2-week treatment, participants are trained in using individualized home practice programs on iPads. They practice approximately daily for six months, checking in weekly with an SLP via videoconferencing software and return for probes monthly. Six months post-treatment testing will take place following completion of the home practice phase and again at 12 months post-treatment.
  Interventions: Behavioral: Intensive Language Action Therapy

INTERVENTIONS:
Behavioral: Intensive Language Action Therapy

SUMMARY:
In this study the investigators are examining the effectiveness of intensive speech therapy in chronic moderate-to-severe stroke-induced aphasia under two conditions - responses "constrained" or unconstrained to speech. Both treatments involve massed practice communicating, using intensive language action therapy 3 hours/day, 5 days/week for two weeks, followed by six months of a home practice program. One treatment stresses spoken responses as the preferred expressive modality during intensive therapy. Before and after treatment, and following the home practice program and a period of no practice, the investigators will administer several tests and discourse samples to examine changes associated with the treatments. Participants will also undergo structural and functional MRI testing at these time points. The investigators will also attempt to quantify the degree to which improvements following intensive language therapy and home practice correlate with changes in Quality of Life measures as perceived by both participants with aphasia and their significant others. It is hypothesized that, whereas both treatments will lead to improvements in naming practiced words and communicating, outcomes will be enhanced for the group randomly assigned to the "constraint" condition. Moreover, performance will be enhanced on words practiced during the home practice program, including those that were not practiced during intensive therapy. Improved naming will correlate with modulation of 'signature' language and attentional networks, whose variability will depend on remaining viable brain structures. Initial severity and site/extent of lesion should predict patients' ability to transfer gains in naming to improvements in discourse.

ELIGIBILITY:
Inclusion Criteria:

* unilateral left hemisphere stroke at least 6 months earlier
* aphasia with moderate-to-severe word retrieval impairments
* at least 21 years of age
* premorbidly right handed
* native speaker of English

Exclusion Criteria:

* history of developmental learning difficulties
* history of prior neurological illnesses
* chronic medical illnesses that restrict participation in intensive therapy
* recent alcohol or drug dependence
* severe uncorrected impairments of vision or hearing
* any contraindication to a 3T MRI procedure (e.g., claustrophobia, metal implants or fragments in body, pregnancy)

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02-26 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-07-09 (Actual)

PRIMARY OUTCOMES:
• Change from baseline on Confrontation Naming Task | Change will be assessed immediately post-treatment (2 weeks)

SECONDARY OUTCOMES:
Change from baseline Boston Diagnostic Aphasia Examination | Change will be assessed immediately post-treatment (2 weeks)

OTHER OUTCOMES:
Change from baseline Boston Naming Test | Change will be assessed immediately post-treatment (2 weeks)
Change from baseline discourse samples | Change will be assessed post-home practice program (approx. 6 months)
Change from baseline Assessment of Living with Aphasia | Change will be assessed post-home practice program (approx. 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacquie Kurland, Ph.D., Principal Investigator — UMass Amherst
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States